CLINICAL TRIAL: NCT06563609
Title: Combined Physical Rehabilitation and Individualized Nutritional Support Versus Standard of Care During In-hospital Endocarditis Treatment
Brief Title: Combined Rehabilitation and Nutritional Support vs. Standard Care in In-Hospital Endocarditis Treatment
Acronym: ENDOCARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Johannes Grand (Other)
Responsible Party: Sponsor-Investigator, Johannes Grand, MD, PhD, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ENDOCARE-001
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Infective Endocarditis; Endocarditis, Bacterial; Infection; Heart; Bacteremia; Cardiac Rehabilitation; Nutrition Intervention; Physical Therapy; Probiotic Intervention
Keywords: Infective endocarditis; Endocarditis team; Physical Therapy; Individualized Nutritional Support; Probiotic yeast Saccharomyces Boulardii; Cardiac rehabilitation
MeSH Terms: conditions — Endocarditis; Endocarditis, Bacterial; Infections; Bacteremia

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, randomized, single-center, 2-by-2 factorial clinical trial with co-enrolment into two different non-pharmacological interventions.
  * A combined Intensive physical Therapy and individualised Nutritional Support intervention and administration of probiotic yeast Saccharomyces boulardii
  * A combined Intensive physical Therapy and individualised Nutritional Support intervention and NO administration of probiotic yeast Saccharomyces boulardii
  * Administration of probiotic yeast Saccharomyces boulardii and NO Intensive physical Therapy and individualised Nutritional Support.
  * NO administration of probiotic yeast Saccharomyces boulardii and NO Intensive physical Therapy and individualised Nutritional Support. Patients will receive standard hospital care
Who Masked: Participant
Masking Description: There are none apart from listen above
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Integrated Physical Therapy and Nutritional Support with Probiotic Saccharomyces boulardii (Active Comparator): Intensive physical therapy + individualised nutritional support + administration of probiotic yeast saccharomyces boulardii
  Interventions: Behavioral: Intensive physical Therapy; Dietary Supplement: Probiotic treatment; Behavioral: Individualised Nutritional Support
- A combined Intensive physical Therapy and individualised Nutritional Support intervention (Active Comparator): Intensive physical Therapy + Individualised Nutritional Support
  Interventions: Behavioral: Intensive physical Therapy; Behavioral: Individualised Nutritional Support
- Administration of probiotic yeast Saccharomyces boulardii (Active Comparator): Administration of probiotic yeast Saccharomyces boulardii
  Interventions: Dietary Supplement: Probiotic treatment
- Control group (Placebo Comparator): Standard hospital care
  Interventions: Other: Standard hospital care

INTERVENTIONS:
Behavioral: Intensive physical Therapy — Tailored exercise programs supervised by trained physiotherapists, focusing on improving cardiorespiratory fitness, strength, and functional capacity.
  Arms: A combined Intensive physical Therapy and individualised Nutritional Support intervention; Integrated Physical Therapy and Nutritional Support with Probiotic Saccharomyces boulardii
Dietary Supplement: Probiotic treatment — Administration of probiotic yeast Saccharomyces boulardii twice daily
  Arms: Administration of probiotic yeast Saccharomyces boulardii; Integrated Physical Therapy and Nutritional Support with Probiotic Saccharomyces boulardii
Behavioral: Individualised Nutritional Support — Personalized nutritional plans guided by a dietitian, addressing malnutrition and caloric/protein deficiencies with daily caloric intake adjustments and supplements if necessary based on the EFFORT trial.
  Arms: A combined Intensive physical Therapy and individualised Nutritional Support intervention; Integrated Physical Therapy and Nutritional Support with Probiotic Saccharomyces boulardii
Other: Standard hospital care — Patients will receive standard hospital care
  Arms: Control group

SUMMARY:
Infective endocarditis (IE) is associated with high morbidity and mortality. Patients with IE are affected by a lengthy hospitalization, leading to physical deconditioning and a rapid decline in physical fitness, muscle mass and strength. Moreover, prolonged antibiotic regimens frequently result in nausea, antibiotic-associated diarrhea and Clostridioides difficile (C.difficile) intestinal infections that further negatively affect patient health. These physical challenges are further exacerbated by the negative impact on mental health, increasing the overall burden of the illness. Implementing a targeted rehabilitative strategy in the hospital setting may therefore improve patient care including physical health and overall quality of life during hospitalization.

DETAILED DESCRIPTION:
BACKGROUND:

Infective endocarditis (IE) is a severe infection of the heart's inner lining, typically the valves, carrying high risks of acute heart failure and death. Patients often face extended hospitalizations (up to six weeks or longer) for intravenous antibiotic treatments, with 30-50% requiring urgent valve surgery. The incidence of IE is 8-10 per 100,000 person-years and rising due to aging populations and increased use of cardiac implantable devices, accounting for 650-700 cases annually in Denmark. Without treatment, mortality is nearly 100%, and with treatment, it ranges from 5-30% during the initial hospitalization, influenced by factors such as infection site, causative agent, age, and comorbidities.

IE significantly impacts patients' health due to prolonged hospitalization. Many experience rapid physical decline, including reduced cardiorespiratory fitness, strength, and overall fitness, caused by bed rest, malnutrition, and limited activity. Recovery is often difficult, with worsening physical, mental, and emotional states. The POET trial found poor self-rated health triples mortality risk. Up to 35% of patients do not return to work, and 65% face readmission within a year. Long hospital stays also increase the need for nursing home care.

Malnutrition is common in IE patients, raising risks of death, illness, and impairment. Acute illness amplifies nutritional deficits, worsening muscle wasting and overall health. The EFFORT trial showed early nutritional support reduces mortality and complications, yet no randomized studies have addressed nutrition in IE patients.

Intravenous antibiotics add distress, often causing nausea, diarrhea, and C. difficile infections. Probiotics like S. boulardii show promise in preventing these side effects.

Cardiac rehabilitation has proven benefits for other heart conditions, improving exercise capacity, quality of life, and reducing readmissions. However, evidence is limited for in-hospital IE rehabilitation. Tailored, supervised programs during hospitalization could address physical and mental health needs, improving overall recovery and quality of life.

PRIMARY AIM:

To investigate the effectiveness of individualized physical rehabilitation and nutritional support designed to reduce physical deconditioning and prevent treatment-related harms thus ultimately improving mental health in patients hospitalized with endocarditis.

HYPOTHESES:

Within a 2-by-2 factorial design, a patient-centered, individualized, and adaptable physical rehabilitation and nutritional plan during lengthy hospitalization will improve mental health more than standard care.

Furthermore, in the same factorial framework, a probiotic supplement during antibiotic-treatment will decrease the rate of antibiotic-associated diarrhea compared to no probiotic supplement.

NUTRITIONAL SUPPORT:

In the intervention group, nutritional screening and support begin within 24 hours of randomization. Individualized nutritional plans are developed based on the NRS 2002 protocol and 2018 international guidelines. A dietitian sets energy requirements using the weight-adjusted Harris-Benedict equation and establishes protein intake targets between 1.2-1.5 g/kg of body weight, adjusting to 0.8 g/kg for patients with acute renal failure.

Patients are screened for risk of refeeding syndrome with routine blood tests, including magnesium, phosphate, and other relevant biomarkers (e.g., bilirubin, creatinine, albumin, electrolytes, etc.). The initial dietary plan includes hospital-provided meals, snacks from an "à la carte" menu, and oral nutritional supplements (ONS). Daily food records monitor intake, and if patients fail to meet 75% of caloric and protein targets for three consecutive days-or earlier based on clinical judgment-escalation to enteral tube feeding or parenteral feeding is initiated.

INDIVIDUALLY PLANNED PHYSICAL EXERCISE BY AN INTERDISCIPLINARY TEAM LEAD BY A SPECIALIZED REHABILITATION PHYSIOTHERAPIST:

The ENDOCARE team, consisting of a cardiologist, nurse, and physiotherapist, optionally involving a family member, will meet with the patient the first weekday after inclusion to design a personalized exercise regimen. This regimen accounts for comorbidities, performance status, disease severity, and support resources. Weekly meetings with the team will address patient concerns and ensure optimal care.

Exercise Modalities

Patients will participate in Intensive Exercise to reduce deconditioning and enhance well-being, focusing on:

Progressive Resistance Exercise: Major muscle groups (e.g., leg presses, arm rows, arm pushes) are targeted with 2-3 sessions/week, using stationary equipment or elastic bands. Training follows a linear progression (3 sets per exercise starting at 15 ± 2 RM, progressing to 10 ± 2 RM) and integrates principles like range of motion and time under tension.

Cardiovascular Exercise: Sessions involve 20 minutes of moderate-intensity exercise (Borg RPE 12-14) 3-4 times/week, using arm ergometers or stationary beds. Intensity and structure (continuous or interval) are adjusted based on patient preference.

Physical Activity Daily physical activity, guided by Danish recommendations (10,000 steps/day), is encouraged using a gradual progression model (e.g., PACE-UP). Activity monitoring is supported by SENS motion accelerometers, with data transferred to a smartphone app. Depending on funding, tablets may provide real-time feedback on activity levels near patient beds.

Control Group Patients in the control group receive standard hospital care, including an initial physiotherapist assessment and 1-2 supervised or self-managed exercise sessions per week.

Risks Potential risks include musculoskeletal injuries (e.g., strains, sprains), fatigue, and overtraining.

GUIDE FOR PROBIOTIC ADMINISTRATION:

In the intervention group, S. boulardii treatment begins at inclusion. Patients will receive Sacchaflor capsules (Pharmaforce Aps), containing S. boulardii (5×10^9 DBVPG 6763 strain) and mannan oligosaccharide (MOS), a supplement derived from Saccharomyces cerevisiae. The capsules are administered twice daily until the end of antibiotic treatment. If the patient is discharged with continued antibiotics, S. boulardii will be used for up to 30 more days.

In the control group, no probiotics will be given for 30 days post inclusion.

Possible side effects include gastrointestinal disturbances (e.g., flatulence, bloating, constipation) and, rarely, fungemia or allergic reactions).

ELIGIBILITY:
INCLUSION CRITERIA

* Clinical diagnosis of left-sided (native, prosthetic, or culture-negative) bacterial infective endocarditis mandating iv antibiotic treatment, including Cardiac Implantable Electronic Devices infections, irrespective of cause and location as defined by the ESC modified Duke Criteria
* Age ≥ 18 years

EXCLUSION CRITERIA

* Hemodynamic instability (defined as a systolic blood pressure <90 mmHg and lactate >2.2 mmol/l measured in an arterial blood gas.
* Expected to be discharged within 3 days
* Immunocompromised due to severe combined immunodeficiency, HIV, or hematological malignancy
* Fungal endocarditis
* Pregnancy
* Unwilling or unable to sign or understand informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-12-07 (Actual); Study Completion 2025-12-07 (Actual)

PRIMARY OUTCOMES:
Mental health (MH) measured by the standardized Short Form 36 (SF-36) | 30 days
  Mental Component Summary (MCS) of the Medical Outcome Study Short Form 36 version 2 (SF-36) which has been validated in Danish and in cardiac populations and is widely used in controlled clinical trials. Scores range from 0 to 100, with higher scores indicating better-perceived health

SECONDARY OUTCOMES:
Change in number of sit and stand in 30 seconds from baseline to 14 days | 14 days
  Sit and stand test
Quality of life from EQ-5D | 14, 30, and 90 days follow-up
  Quality of life measured efte 30 days using EuroQol-5 Domain (EQ-5D) The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Days alive without diarrhea | 30 days in hospital and 90 days out of hospital
  Assessment with Bristol Stool Chart
Days alive and out of hospital | 30 day in hospital, and 90 day out-of-hospital
All-cause mortality | 30 days

OTHER OUTCOMES:
Albumin Measurement | 14 days
  Blood test
The occurrence of C. difficile infection | 14 days and 30 days
  Defined as an episode of diarrhea combined with the detection of toxins A or B, or both, from a rectal swap
NT-proBNP | 14 days after admission
  Blood test
Left ventricular ejection fraction | 14 days
  Left ventricular ejection fraction measured with echocardiography
SENS motion | First 7 days
  Number of daily steps
Self-rated Hospital Anxiety and Depression Scale (HAD) | 14, 30, and 90 days follow-up
  The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depressio
HbA1c | Day 14
  Blood test
Lipids | Day 14
  Blood test
Number of patients at risk of malnutrition | Day 14
Number of patients getting daily average of at least 75% of the caloric and protein targets on day 4 | Day 14
Number of patients required for enteral tube feeding or parenteral feeding | Day 14
Grip strength | 14, 30, and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Grand, MD, PhD, Principal Investigator — Copenhagen University Hospital Amager-Hvidovre, Department of Cardiology
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the publication will be shared. Data will be available beginning after publicatoin of the main papers. Access will be granted to researchers who provide a methodologically sound proposal, which will be reviewed by the national governing body for approval both regarding ethics and patients data safety.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1/1 2028 - 31/12 2037
Access Criteria: Access will be granted to researchers who provide a methodologically sound proposal. All data avaiable will potentially be shared if approved be athorities. Data transfer can be made through an approoved data transfar system, which should be made available by the researcher seeking the data.